CLINICAL TRIAL: NCT02464410
Title: Primary Care Intervention to Reduce Prescription Opioid Overdoses
Acronym: POST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 13-322
Record Dates: First submitted 2015-05-21; First posted 2015-06-08 (Estimated); Results first posted 2022-09-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pain; Drug Overdose; Opioid Use Disorders
Keywords: Opioid analgesics; Primary care; Veterans; Motivational interviewing; Cognitive behavioral therapy; Self-efficacy; Behavioral symptoms; Injuries; Opioid Safety
MeSH Terms: conditions — Pain; Drug Overdose; Opioid-Related Disorders; Behavioral Symptoms; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Intervention (Experimental): The intervention session combines elements of motivational enhancement (ME) and cognitive behavioral therapy (CBT) and uses the structure of ME brief interventions. The motivational session is overlaid on the VA long-term opioid therapy informed consent process.
  Interventions: Behavioral: Motivational intervention; Other: Long-term opioid therapy informed consent
- Enhanced Usual Care (Active Comparator): In addition to covering the VHA's long-term OA informed consent process, the enhanced usual care (EUC) condition provides educational content related to the biology of pain response and an overview of pain conditions. The overall style is didactic. This EUC condition will include some information related to risks of opioid use as part of the informed consent and will consequently have sufficient face validity as an intervention on opioid safety to effectively blind participant to randomization. However, the EUC therapist will not use the motivational enhancement approach of discussing strategies for avoiding these risks. It is designed to be equal in length to the motivational intervention.
  Interventions: Behavioral: Psycho-educational control; Other: Long-term opioid therapy informed consent

INTERVENTIONS:
Behavioral: Motivational intervention — The intervention session combines elements of motivational enhancement (ME) and cognitive behavioral therapy (CBT). Similar to other ME brief interventions, the intervention content will be covered in a single session. Participants are presented with a variety of risk reduction strategies and strategies for coping with pain that may reduce reliance on opioids for managing pain.
  Arms: Motivational Intervention
Behavioral: Psycho-educational control — The educational control condition provides educational content related to the biology of pain response and an overview of pain conditions. The overall style is didactic.
  Arms: Enhanced Usual Care
Other: Long-term opioid therapy informed consent — The Veterans Health Administration instituted a requirement that all patients receiving long-term opioid therapy receive an informed consent process that reviews the risks of opioid therapy. All individuals eligible for this study will meet this definition of long-term opioid therapy. The study therapists for both study arms will deliver the informed consent process during the sessions as part of treatment as usual.

SUMMARY:
The high rate of adverse events, including overdose, resulting from opioid pain medication use threatens the quality and safety of pain care in the Veterans Health Administration (VHA) and elsewhere and is a critical public health problem in the United States. Pain is a highly common condition among VHA patients, and opioid therapy constitutes a primary mode of pain treatment.

This study seeks to address this issue by conducting a randomized controlled trial of a brief conversation to improve opioid safety among Veteran patients receiving long-term opioid therapy. Veterans receiving opioid therapy for pain in primary care will be recruited and randomized to receive either a single session motivational intervention focused on safe opioid use or an equal attention control condition. The primary hypothesis is that the motivational intervention will improve opioid safety, decrease risk behaviors, aberrant opioid use, and total quantities of opioids prescribed relative to the control condition. Study findings will inform efforts to ensure the safety and well-being of Veteran patients with pain.

DETAILED DESCRIPTION:
Adverse outcomes, including overdose, related to opioid use have increased and represent a significant threat to the safety and quality of VHA pain care as well as a national public health concern. Efforts are underway to change opioid prescribing behavior, but concurrent strategies are needed to address patient behaviors that decrease opioid safety and thus increase opioid overdose risk. Overdoses result from a range of behaviors, including taking more than prescribed, using multiple substances with synergistic effects, and injecting/snorting crushed pills to get high. Factors such as having a mental health condition have been found to increase risk of overdose among Veterans receiving opioids for pain. Given the range of risk behaviors and relevant patient factors, tailored opioid risk reduction strategies are urgently needed. Motivational enhancement (ME) is an evidence-based strategy that uses tailoring to enact behavior change through improving self-efficacy and motivation. Recent VHA initiatives to increase behavioral health providers in primary care, such as Primary Care-Mental Health Integration (PC-MHI), provide a clear opportunity to deliver ME interventions to the many patients treated for long-term pain in primary care. Although the impact of ME on overdose risk behavior is unknown, the use of an ME approach to improve opioid safety and reduce risk behaviors is potentially well-suited to the context of long-term opioid pain care, when total and immediate discontinuation of opioid use is often unfeasible.

The proposed Prescription Opioid Safety Trial (POST) study will be a randomized controlled trial of a brief, tailored ME conversation that incorporates cognitive behavioral strategies to increase pain coping and is aimed at improving patients' opioid safety. The study will recruit 450 patients from primary care clinics at the VA Ann Arbor Healthcare System. Patients with long-term opioid use, defined as treatment for at least 84 days covered within the last 90 days, who are prescribed opioid doses of 20 morphine-equivalent mg/day or greater (an indicator of overdose risk) will be screened and recruited into the study. Participants will then be randomized to either the intervention (n = 225) or an enhanced usual care (EUC) condition (n = 225). Pharmacy records and patient self-report will be assessed at baseline and 3-, 6-, and 12-month follow-ups to measure key outcomes.

The specific aims are:

Aim 1) to examine if patients randomly assigned to a brief opioid safety intervention report reduced overdose risk behaviors (e.g., higher dose, concurrent alcohol use, concurrent other drug/medication use, returning to normal dose after breaks in use) over one year of follow-up compared to patients assigned to equal attention EUC.

Aim 2) to examine if patients randomly assigned to a brief opioid safety intervention have lower total quantities of opioids prescribed (from pharmacy fill records) and aberrant opioid use (e.g., using for reasons other than pain, obtaining opioids from someone other than primary provider) over one year of follow-up compared to patients assigned to equal attention EUC.

The study has two secondary aims: 1) to examine if patients randomly assigned to the brief intervention have fewer non-fatal overdoses and other medication-related adverse events (emergency department visits, over-sedation, injuries), better functioning, and more often store and dispose of opioids safely compared to patients assigned to EUC; and 2) to examine mediators (motivation and self-efficacy) and moderators (OIF/OEF/OND status, baseline mental health) of intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Ann Arbor VA Medical Center receiving treatment in a primary care clinic
* Currently prescribed 20 morphine-equivalent mg (MEM) per day or more of an opioid
* Received opioid therapy for at least 90 days
* 18 years of age or older

Exclusion Criteria:

* Plans to stop opioids or reduce dose to below 20 MEM/day in the next 6 months
* Use of fentanyl, due to the difficulty in determining morphine equivalency
* A terminal cancer diagnosis
* Acute suicidality requiring immediate treatment
* Moderately severe cognitive impairment
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Bohnert, PhD MHS BA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Humphreys K, Shover CL, Andrews CM, Bohnert ASB, Brandeau ML, Caulkins JP, Chen JH, Cuellar MF, Hurd YL, Juurlink DN, Koh HK, Krebs EE, Lembke A, Mackey SC, Larrimore Ouellette L, Suffoletto B, Timko C. Responding to the opioid crisis in North America and beyond: recommendations of the Stanford-Lancet Commission. Lancet. 2022 Feb 5;399(10324):555-604. doi: 10.1016/S0140-6736(21)02252-2. Epub 2022 Feb 2. No abstract available. PMID 35122753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Intervention | Enhanced Usual Care
Started | 147 | 152
3-month Follow-up | 137 | 138
6-month Follow-up | 132 | 140
12-month Follow-up | 125 | 136
Completed | 125 | 136
Not Completed | 22 | 16
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 7 | 9
Not completed — Withdrawal by Subject | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 147 | 152 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 87 | 155
  >=65 years | 79 | 65 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 132 | 144 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 141 | 150 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 125 | 125 | 250
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 147 | 152 | 299
Overdose risk behaviors [Mean (Standard Deviation); unit: units on a scale] — This scale is a total sum of 9 items assessing participant's self-report of engaging in behavior that increases risk for overdose. Higher scores indicate greater risk for overdose. The range for this measure is 0 to 9 in one assessment.
  units on a scale | 1.63 (1.16) | 1.75 (1.26) | 1.69 (1.21)
Aberrant opioid use [Mean (Standard Deviation); unit: units on a scale] — This measure contained 8 items from the Current Opioid Misuse Measure. Items were assessed on a scale of "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)." A sum score took a range of 0 to 32, with higher numbers indicating more non-medical opioid use. Population: The number of participants analyzed are adjusted for missing data.
  units on a scale
    number analyzed (Participants) | 146 | 152 | 298
    (all) | 4.16 (3.58) | 3.77 (3.43) | 3.96 (3.51)
Average number of days prescribed opioid use based on pharmacy records [Mean (Standard Deviation); unit: Days of Prescribed Opioid Use] — Number of days prescribed opioid use was pulled from pharmacy records. For follow-up periods, times no dose were included to create averages over periods. Patients without medications during their follow-up period were included with a dose of zero.
  Days of Prescribed Opioid Use | 51.57 (39.75) | 47.54 (38.96) | 49.52 (39.34)
Participants with non-fatal overdose experiences [Number; unit: Number with Overdose Experiences] — This scale is the number of overdose experiences as self-reported in the Overdose Experiences questionnaire. This item is the number of participants whom endorsed having experienced an overdose at that time period. Population: The number of participants analyzed are adjusted for missing data
  Number with Overdose Experiences
    number analyzed (Participants) | 147 | 149 | 296
    (all) | 29 | 29 | 58
Treatment utilization [Mean (Standard Deviation); unit: Number of Visits to the Emergency Dept] — Number of visits to the emergency department, for medical, mental health or substance use visits, across VA and non-VA hospitals from the Treatment Service Utilization Questionnaire. The numbers reported are the mean number of visits among those participants that had any emergency department visits at each time point. Population: Due to lost to follow-up, death, participant withdrawal, or the lack of visits to the emergency department, the number analyzed varied throughout the study.
  Number of Visits to the Emergency Dept
    number analyzed (Participants) | 81 | 75 | 156
    (all) | 1.29 (1.68) | 1.28 (1.98) | 1.28 (1.83)
Other (non-overdose) injuries from the Revised Injury Behavior Checklist Questionnaire [Count of Participants; unit: Participants] — This scale is the number of non-overdose injuries assessed through the Revised Injury Behavior Checklist questionnaire, focusing on 4 topics (Injury 1. by violence or by being physically attacked; 2. By falling; 3. By a motor vehicle or by being hit by a moving vehicle while walking; 4. While riding a bicycle, skateboard, or rollerblading). This item is a count of participants who responded that they were injured during any of these types of activities and received treatment. Population: The number of participants analyzed are adjusted for missing data.
  Participants
    number analyzed (Participants) | 146 | 151 | 297
    (all) | 18 | 13 | 31
Scores on an opioid storage and disposal knowledge and behaviors questionnaire [Mean (Standard Deviation); unit: units on a scale] — This scale assesses safe storage and disposal of prescription opioid medications with 6 items. Items were assessed on a scale of "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)." A sum score took a range of 0 to 24, with higher numbers indicating less safe practices. The sum of the score of the 6 items was used to find the mean scores for those in each arm.
  units on a scale | 1.4 (1.78) | 1.16 (1.91) | 1.28 (1.85)
Level of oversedation as an opioid side effect [Mean (Standard Deviation); unit: units on a scale] — The level of oversedation as an opioid side effect was assessed using two items from the Pain Treatment Satisfaction Scale looking at side effects of opioid medications (excessive fatigue and drowsiness). Items were assessed on a scale of 0 (did not experience) to 5 (extremely bothered). A sum score ranged from 0 to 10 with a higher score indicating the potential for more oversedation. Population: The numbers of participants analyzed are adjusted for missing data.
  units on a scale
    number analyzed (Participants) | 142 | 147 | 289
    (all) | 2.80 (2.55) | 2.29 (2.45) | 2.54 (2.51)
General physical and mental functioning from Veteran Short Form questionnaire scores [Mean (Standard Deviation); unit: units on a scale] — A modified Veterans RAND 12-item health survey was used to assess general health. One item was scored from 1 (Excellent) to 5 (Poor). Score means were compared at baseline and each follow-up. Population: The number of participants analyzed are adjusted for missing data.
  units on a scale
    number analyzed (Participants) | 147 | 151 | 298
    (all) | 3.49 (0.95) | 3.62 (0.98) | 3.55 (0.96)
Pain-specific disability score [Mean (Standard Deviation); unit: units on a scale] — This scale is a sub-section of the Brief Pain Inventory that assesses the impact of pain on functioning across 7 different activities. Activities are assessed on a Likert scale from "Does not interfere (0)" to "Completely interferes (10)". BPI pain interference was scored as the mean of the seven interference items, scores range from 0 to 10, with a mean score of 10 (maximum score) indicating a complete interference in all activities. Population: The number of participants analyzed are adjusted for missing data.
  units on a scale
    number analyzed (Participants) | 147 | 151 | 298
    (all) | 5.19 (2.70) | 5.55 (2.54) | 5.38 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: Overdose Risk Behaviors
Description: This scale is a total sum of 9 items assessing participant's self-report of engaging in behavior that increases risk for overdose. Higher scores indicate greater risk for overdose. The range for this measure is 0 to 9 in one assessment.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: Due to lost to follow-up, death, missing data, or participant withdrawal, the number analyzed varied throughout the follow-up periods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 137 | 138
  3-Month Follow-up | 1.31 (1.14) | 1.21 (1.09)
  6-Month Follow-up: number analyzed (Participants) | 131 | 140
  6-Month Follow-up | 1.45 (1.20) | 1.25 (1.29)
  12-Month Follow-up: number analyzed (Participants) | 125 | 136
  12-Month Follow-up | 1.38 (1.29) | 1.07 (1.05)

2. Primary Outcome: Aberrant Opioid Use
Description: This measure contained 8 self-reported items from the Current Opioid Misuse Measure. Items were assessed on a scale of "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)." A sum score took a range of 0 to 32, with higher numbers indicating more non-medical opioid use.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 137 | 137
  3-Month Follow-up | 2.95 (3.04) | 2.51 (2.74)
  6-Month Follow-up: number analyzed (Participants) | 131 | 140
  6-Month Follow-up | 2.87 (3.06) | 2.68 (3.11)
  12-Month Follow-up: number analyzed (Participants) | 123 | 134
  12-Month Follow-up | 2.80 (3.08) | 2.73 (3.35)

3. Primary Outcome: Average Number of Days Prescribed Opioid Use Based on Pharmacy Records
Description: Number of days prescribed opioid use was pulled from pharmacy records. For follow-up periods, times no dose were included to create averages over periods. Patients without medications during their follow-up period were included with a dose of zero.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: All participants were included in this analysis as this was taken from Electronic Health Records and did not rely on follow-up survey responses.
Measure: Mean (Standard Deviation); unit: Days of Prescribed Opioid Use
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 147 | 152
Days of Prescribed Opioid Use
  3-Month Follow-up | 48.23 (38.97) | 45.81 (41.06)
  6-Month Follow-up | 44.75 (38.70) | 42.54 (41.08)
  12-Month Follow-up | 42.19 (38.92) | 37.56 (38.83)

4. Secondary Outcome: Number of Participants With Non-fatal Overdose Experiences
Description: This scale is the number of overdose experiences as self-reported in the Overdose Experiences questionnaire. This item is a number of participants whom endorsed having experienced an overdose at that time period.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: Due to lost to follow-up, death, missing data, or participant withdrawal, the number analyzed varied throughout the follow-up periods. The Overall Number of Participants Analyzed includes participants with at least one outcome assessment at each timepoint.
Measure: Number; unit: participants with OD
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
participants with OD
  3-Month Follow-up: number analyzed (Participants) | 136 | 138
  3-Month Follow-up | 1 | 0
  6-Month Follow-up: number analyzed (Participants) | 131 | 140
  6-Month Follow-up | 2 | 1
  12-Month Follow-up: number analyzed (Participants) | 124 | 136
  12-Month Follow-up | 0 | 1

5. Secondary Outcome: Treatment Utilization
Description: Number of visits to the emergency department, for medical, mental health or substance use visits, across VA and non-VA hospitals from the Treatment Service Utilization Questionnaire. The numbers reported are the mean number of visits among those participants that had any emergency department visits at each time point.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: Due to lost to follow-up, death, missing data, participant withdrawal, or the lack of visits to the emergency department, the number analyzed varied throughout the study.
Measure: Mean (Standard Deviation); unit: Visits to the Emergency Dept
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
Visits to the Emergency Dept
  3-Month Follow-up: number analyzed (Participants) | 28 | 36
  3-Month Follow-up | 1.50 (0.84) | 1.81 (1.24)
  6-Month Follow-up: number analyzed (Participants) | 28 | 27
  6-Month Follow-up | 1.61 (1.77) | 2.11 (2.31)
  12-Month Follow-up: number analyzed (Participants) | 40 | 47
  12-Month Follow-up | 2.20 (3.27) | 2.04 (1.85)

6. Secondary Outcome: Other (Non-overdose) Injuries From the Revised Injury Behavior Checklist Questionnaire
Description: This scale is the number of non-overdose injuries assessed through the Revised Injury Behavior Checklist questionnaire, focusing on 4 topics (Injury 1. by violence or by being physically attacked; 2. By falling; 3. By a motor vehicle or by being hit by a moving vehicle while walking; 4. While riding a bicycle, skateboard, or rollerblading). This item is a count of participants who responded that they were injured during any of these types of activities and received treatment.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
Participants
  3-Month Follow-up: number analyzed (Participants) | 137 | 138
  3-Month Follow-up | 5 | 4
  6-Month Follow-up: number analyzed (Participants) | 131 | 140
  6-Month Follow-up | 4 | 5
  12-Month Follow-up: number analyzed (Participants) | 125 | 136
  12-Month Follow-up | 11 | 4

7. Secondary Outcome: Scores on an Opioid Storage and Disposal Knowledge and Behaviors Questionnaire
Description: This scale assesses safe storage and disposal of prescription opioid medications with 6 items. Items were assessed on a scale of "never (0)," "rarely (1)," "sometimes (2)," "often (3)," and "very often (4)." A sum score took a range of 0 to 24, with higher numbers indicating less safe practices. The sum of the score of the 6 items was used to find the mean scores for those in each arm.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 137 | 138
  3-Month Follow-up | 0.95 (1.47) | 0.68 (1.28)
  6-Month Follow-up: number analyzed (Participants) | 131 | 140
  6-Month Follow-up | 1.07 (1.63) | 0.69 (1.37)
  12-Month Follow-up: number analyzed (Participants) | 124 | 136
  12-Month Follow-up | 1.13 (1.82) | 0.76 (1.45)

8. Secondary Outcome: Level of Oversedation as an Opioid Side Effect
Description: The level of oversedation as an opioid side effect was assessed using two items from the Pain Treatment Satisfaction Scale looking at side effects of opioid medications (excessive fatigue and drowsiness). Items were assessed on a scale of 0 (did not experience) to 5 (extremely bothered). A sum score ranged from 0 to 10 with a higher score indicating the potential for more oversedation.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 135 | 138
  3-Month Follow-up | 1.66 (2.20) | 1.96 (2.59)
  6-Month Follow-up: number analyzed (Participants) | 129 | 138
  6-Month Follow-up | 1.57 (2.05) | 2.08 (2.55)
  12-Month Follow-up: number analyzed (Participants) | 123 | 129
  12-Month Follow-up | 2.36 (2.46) | 2.25 (2.59)

9. Secondary Outcome: General Physical and Mental Functioning From Short Form-12 Questionnaire Scores
Description: A modified Veterans RAND 12-item health survey was used to assess general health. One item was scored from 1 (Excellent) to 5 (Poor). Score means were compared at baseline and each follow-up.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 136 | 138
  3-Month Follow-up | 3.57 (0.89) | 3.70 (0.95)
  6-Month Follow-up: number analyzed (Participants) | 130 | 139
  6-Month Follow-up | 3.63 (0.94) | 3.76 (0.99)
  12-Month Follow-up: number analyzed (Participants) | 125 | 135
  12-Month Follow-up | 3.71 (0.81) | 3.79 (0.93)

10. Secondary Outcome: Pain-specific Disability Score From an Adapted Version of Brief Pain Inventory Questionnaire
Description: This scale is a sub-section of the Brief Pain Inventory that assesses the impact of pain on functioning across 7 different activities. Activities are assessed on a Likert scale from "Does not interfere (0)" to "Completely interferes (10)". BPI pain interference was scored as the mean of the seven interference items, scores range from 0 to 10, with a mean score of 10 (maximum score) indicating a complete interference in all activities.
Time Frame: 3-, 6-, and 12-months post-baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Intervention | Enhanced Usual Care
Number analyzed (Participants) | 137 | 140
score on a scale
  3-Month Follow-up: number analyzed (Participants) | 136 | 137
  3-Month Follow-up | 4.86 (2.87) | 5.10 (4.64)
  6-Month Follow-up: number analyzed (Participants) | 129 | 139
  6-Month Follow-up | 4.89 (2.66) | 5.16 (2.88)
  12-Month Follow-up: number analyzed (Participants) | 125 | 135
  12-Month Follow-up | 4.89 (4.40) | 5.41 (2.51)

ADVERSE EVENTS:
Time Frame: Collected over 12 months post-baseline assessment
Description: Adverse events were discovered while completing retention activities, such as EHR checks or calling and talking to family members. All participants were at risk of all-cause mortality, or some unanticipated serious adverse event.
Arm/Group | Motivational Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 3/147 | 4/152
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/152
Other Adverse Events (participants affected / at risk) | 0/147 | 0/152

LIMITATIONS AND CAVEATS:
During the course of this project, the VA changed their opioid prescribing practices in response to the Opioid Safety Initiative. This changed the potential participants for this study (patients prescribed more than 50 MEM), so we updated our enrollment criteria to 20 MEM. We still did not meet our enrollment goal as we had reached saturation of the potential participant pool of patients in primary care at the local VA hospital. At the same time, our overall retention rate is 87.3%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT02464410/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT02464410/ICF_001.pdf